CLINICAL TRIAL: NCT05208385
Title: Effectiveness of the Video-assisted Umbilical Fascial Closure in Laparoscopic Cholecystectomy: Prospective Randomized Clinical Trial of 240 Patients
Brief Title: Video-assisted Umbilical Fascial Closure in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Elif Colak, Associate Professor, Samsun Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KAEK2020/3 /1
Record Dates: First submitted 2021-12-27; First posted 2022-01-26 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cholelithiasis (Without Cholecystitis); Pain, Postoperative; Hernia Incisional
Keywords: laparoscopic cholecystectomy; pain; trocar site hernia
MeSH Terms: conditions — Cholelithiasis; Pain, Postoperative; Incisional Hernia; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard umbilical trocar incision closure (UC) (Other): standard umbilical trocar incision closure
  Interventions: Procedure: video-assisted umbilical closure
- Video-assisted umbilical trocar incision closure (UCVA)) (Active Comparator): video-assisted umbilical trocar incision closure
  Interventions: Procedure: video-assisted umbilical closure

INTERVENTIONS:
Procedure: video-assisted umbilical closure — video-assisted umbilical closure
  Other Names: standard umbilical fascial closure

SUMMARY:
A prospective randomized study was performed including consecutive patients who underwent an elective laparoscopic cholecystectomy (LC) for symptomatic cholelithiasis during the 18 months period. This prospective randomized trial aims to compare two umbilical closure techniques for trocar site hernia (TSH) in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is currently the gold standard in the treatment for symptomatic cholelithiasis that offers a variety of advantages over conventional open surgery such as shorter recovery time, better cosmesis, less wound complication rates, and less pain (1,2). Despite these advantages, LC can result in unique complications. Among these complications, trocar site hernia (TSH) is one of the most important complications because laparoscopic cholecystectomy promises smaller abdominal incisions and better cosmetic outcomes. A second surgical intervention due to TSH may overshadow the gains of the previous laparoscopic surgery. In studies conducted to date, the rate of trocar hernia in laparoscopic cholecystectomy has been presented at very different rates. Many studies have shown that the most frequent site of TSH is the umbilical trocar site (3-6).

To avoid this important complication of laparoscopic cholecystectomy, many different techniques have been described to date for trocar port fascia repair (7-12). Most of these techniques require special devices. In addition, a few studies compare these techniques with standard fascial closure, which is mostly used by surgeons (11,12).

We hypothesized that the fascial closure of the umbilical trocar incision under the intra-abdominal vision with the laparoscopic camera could be reduced TSH. This prospective randomized controlled study aims to assess whether fascial closure of umbilical trocar site under direct laparoscopic vision in LC can reduce the incidence of TSH.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* symptomatic cholelithiasis

Exclusion Criteria:

* acute cholecystitis
* age under 18 years
* previous umbilical hernia repair
* pre-existing umbilical hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Trocar site hernia (TSH) | 18 months
  trocar site hernia presence

SECONDARY OUTCOMES:
Wound infection (WI) | three weeks later
  wound infection
Hematoma (H) | 18 months (postoperative first day and three weeks later)
  Hematoma
Length of hospital stay (LOH) | 18 months
  length of hospital stay (day)
Abdominal Pain | Preoperative first day, postoperative first day
  Abdominal pain assessment by visual analog scale (0 minimum-10 maximum values, higher scores mean worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Elif Colak, Principal Investigator — Samsun Education and Research Hospital
Locations (1):
- Samsun Education and Research Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during the current study are available.
Supporting Information: Study Protocol
Time Frame: January 2021
Access Criteria: The datasets generated during the current study are available.

REFERENCES:
- [Background] Coccolini F, Catena F, Pisano M, Gheza F, Fagiuoli S, Di Saverio S, Leandro G, Montori G, Ceresoli M, Corbella D, Sartelli M, Sugrue M, Ansaloni L. Open versus laparoscopic cholecystectomy in acute cholecystitis. Systematic review and meta-analysis. Int J Surg. 2015 Jun;18:196-204. doi: 10.1016/j.ijsu.2015.04.083. Epub 2015 May 6. PMID 25958296
- [Background] Sanford DE. An Update on Technical Aspects of Cholecystectomy. Surg Clin North Am. 2019 Apr;99(2):245-258. doi: 10.1016/j.suc.2018.11.005. Epub 2019 Feb 10. PMID 30846033
- [Background] Nofal MN, Yousef AJ, Hamdan FF, Oudat AH. Characteristics of Trocar Site Hernia after Laparoscopic Cholecystectomy. Sci Rep. 2020 Feb 18;10(1):2868. doi: 10.1038/s41598-020-59721-w. PMID 32071382
- [Background] Bunting DM. Port-site hernia following laparoscopic cholecystectomy. JSLS. 2010 Oct-Dec;14(4):490-7. doi: 10.4293/108680810X12924466007728. PMID 21605509
- [Background] Erdas E, Dazzi C, Secchi F, Aresu S, Pitzalis A, Barbarossa M, Garau A, Murgia A, Contu P, Licheri S, Pomata M, Farina G. Incidence and risk factors for trocar site hernia following laparoscopic cholecystectomy: a long-term follow-up study. Hernia. 2012 Aug;16(4):431-7. doi: 10.1007/s10029-012-0929-y. Epub 2012 Jun 20. PMID 22714582
- [Background] Comajuncosas J, Hermoso J, Gris P, Jimeno J, Orbeal R, Vallverdu H, Lopez Negre JL, Urgelles J, Estalella L, Pares D. Risk factors for umbilical trocar site incisional hernia in laparoscopic cholecystectomy: a prospective 3-year follow-up study. Am J Surg. 2014 Jan;207(1):1-6. doi: 10.1016/j.amjsurg.2013.05.010. Epub 2013 Oct 7. PMID 24112669
- [Background] Kawai H, Misawa T, Sasaya K, Aoyama Y. Dual-hemostat port closure technique with customized surgical suture after laparoscopic cholecystectomy: Single-center experience. Asian J Endosc Surg. 2020 Jan;13(1):83-88. doi: 10.1111/ases.12690. Epub 2019 Jan 27. PMID 30688041
- [Background] Lasheen AE, Safwat K, Elsheweal A, Ibrahim A, Mahmoud R, Alkilany M, Ismaeil A. Effective, simple, easy procedure for laparoscopic port closure in difficult cases. Ann Med Surg (Lond). 2016 Jul 19;10:36-40. doi: 10.1016/j.amsu.2016.06.014. eCollection 2016 Sep. PMID 27536351
- [Background] Rajendiran A, Maruthupandian D, Karunakaran K, Syed MN. Aneurysm Needle as an Effective Tool in Laparoscopic Port Closure. J Laparoendosc Adv Surg Tech A. 2015 Sep;25(9):744-6. doi: 10.1089/lap.2015.0249. Epub 2015 Aug 19. PMID 26287316
- [Background] Lasheen A, Safwat K, Fiad A, Elmoregy A, Hamed AW. Port-site closure using a modified aptos needle. JSLS. 2013 Apr-Jun;17(2):312-5. doi: 10.4293/108680813X13693422522277. PMID 23925027
- [Background] Calik A, Yucel Y, Topaloglu S, Hos G, Aktas A, Piskin B. Umbilical trocar site closure with Berci's needle after laparoscopic cholecystectomy. Hepatogastroenterology. 2008 Nov-Dec;55(88):1958-61. PMID 19260458
- [Background] Armananzas L, Ruiz-Tovar J, Arroyo A, Garcia-Peche P, Armananzas E, Diez M, Galindo I, Calpena R. Prophylactic mesh vs suture in the closure of the umbilical trocar site after laparoscopic cholecystectomy in high-risk patients for incisional hernia. A randomized clinical trial. J Am Coll Surg. 2014 May;218(5):960-8. doi: 10.1016/j.jamcollsurg.2014.01.049. Epub 2014 Feb 18. PMID 24680572

DOCUMENTS (1):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT05208385/Prot_000.pdf